CLINICAL TRIAL: NCT05120258
Title: Subclavian / Infraclavicular Axillary Vein Collapsibility Index in Pregnant Patients
Brief Title: Can Subclavian / Infraclavicular Axillary Vein Collapsibility Index Predict Post-Spinal Hypotension in Caesarean Section Operations?
Acronym: Cesarean
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, EMİNE ASLANLAR, Assistant professor, Selcuk University
Other Study IDs: SCV
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Post Spinal Hypotension
Keywords: post spinal hypotension, the subclavian vein or infraclavicular axillary vein collapsibility index

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postspinal hypotension (PSH) is a common side effect with an incidence of 15.3% to 33%, which may result in organ hypoperfusion and ischemic events (1,2). In pregnant patients, this incidence may increase to 70% and severe PSH may increase the risk of maternal and fetal complications (3). Therefore, it is important for anesthesiologists to estimate the incidence of PSH in cesarean sections and to identify possible mechanisms (4).

One of the important factors affecting the susceptibility of patients to intraoperative hypotension is the preoperative intravascular volume status. Recently, ultrasonography of the central veins has been used frequently by anesthesiologists in the preoperative period in order to evaluate the intravascular volume status (5). Salama and Elkashlan stated that the collapsibility index of the inferior vena cava is a new predictive value for PSH (6). Choi et al. showed that the subclavian vein or infraclavicular axillary vein collapsibility index is an important predictive value for hypotension after induction of general anesthesia (7).

In this study, we wanted to investigate whether the subclavian vein or infraclavicular axillary vein collapsibility index can be used as a predictive value for PSH in cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Spinal anesthesia
* ceserean operation
* American Society of Anesthesiologists' (ASA) physical status I-II

Exclusion Criteria:

* Patients who underwent cesarean section in emergency conditions
* Patients who underwent cesarean section under general anesthesia
* American Society of Anesthesiologists' (ASA) physical status III-IV

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: ASA I-II physical status patients scheduled for cesarean section under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-08 (Estimated); Primary Completion 2022-01-24 (Estimated); Study Completion 2022-03-02 (Estimated)

PRIMARY OUTCOMES:
Predictive value of Subclavian / Infraclavicular Axillary Vein Collapsibility Index for detecting Postspinal hypotension | 45 min
  Postspinal hypotension (PSH) is a common side effect with an incidence of 15.3 to 33% that may result in organ hypoperfusion and ischaemic events. This incidence is higher in pregnant women with a rate of 70%. Measurement of the IVC diameter and its collapsibility index before spinal anaesthesia has been shown to be a good predictive value of the occurrence of PSH. A previous study showed an acceptable correlation between the collapsibility of SCV (SCV-CI) and collapsibility of IVC (IVC-CI) in surgical and intensive care patients. In this study, we measured the preoperative collapsibility index of the SCV or the infraclavicular axillary vein during respiratory variation, and then examined whether these parameters could predict hypotension after spinal anaesthesia in patients undergoing ceserean

CONTACTS AND LOCATIONS:
Overall Officials: Emine ASLANLAR, assis. prof., Principal Investigator — selcuk univercity medical faculty